CLINICAL TRIAL: NCT02262039
Title: Reducing Operative and Post-operative Morbidity in Living Kidney Donors With the Airseal System: A Randomized Control Trial
Brief Title: Reducing Operative and Post-operative Morbidity in Living Kidney Donors With the Airseal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1405013985
Record Dates: First submitted 2014-07-09; First posted 2014-10-10 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: living; kidney; donors
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Pressure (Active Comparator): Conventional Insufflation with 15mmHg target pressure
  Interventions: Device: Conventional pressure
- Low Pressure (VTI) (Experimental): Valveless recirculating insufflation (VTI) with 10mmHg target pressure
  Interventions: Device: Valveless recirculating insufflation (VTI)

INTERVENTIONS:
Device: Valveless recirculating insufflation (VTI) — 10 mmHg target pressure
  Arms: Low Pressure (VTI)
Device: Conventional pressure — 15 mmHg target pressure
  Arms: Conventional Pressure

SUMMARY:
The purpose of this study is to determine if the Airseal System will reduce post-operative pain and reduce the need for narcotics in laparoscopic living kidney donor surgeries.

DETAILED DESCRIPTION:
Our hypothesis is that Airseal Insufflation System will provide reduced mean operative insufflation pressure and operative mean ETCO2, resulting in improved post-operative pain control and improved operative safety.

The Airseal System has demonstrated decreased variability in intra-abdominal pressure, less post-operative shoulder pain, lower mean ETCO2 and reduced narcotic pain administration. These metrics have been demonstrated in human subjects undergoing gynecologic, urologic and bariatric procedures. The established benefits in a human model provide a foundation for translating this technology to living kidney donors. The advantage lies in the ability to improve pain-related outcomes in this population, which translates into increased living donation; the single solution to reduce mortality for patients suffering from end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Any living donor who has been approved to donate a kidney is eligible to participate.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kulkarni, MD, Study Director — Yale University
Locations (1):
- Yale New Haven Transplantation Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Pressure: 15mmHg target pressure
- Low Pressure (VTI): 10mmHg target pressure
  VTI = Valveless recirculating insufflation
Period: Overall Study
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Started | 14 | 27
Completed | 14 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who agreed to participate completed the study and are included in the analysis.
Groups:
- Low Pressure (VTI): 10mmHg target pressure
  VTI= Valveless recirculating insufflation
- Total: Total of all reporting groups
Arm/Group | Conventional Pressure | Low Pressure (VTI) | Total
Number analyzed (Participants) | 14 | 27 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.3) | 51.6 (14.5) | 47.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 6 | 11 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11 | 22 | 33
  African American | 2 | 2 | 4
  Hispanic | 1 | 3 | 4
Nephrectomy Laterality [Number; unit: participants] — This refers to the location (left side vs. right side) of the kidney removed during the donor surgery
  participants
    Left | 11 | 24 | 35
    Right | 3 | 3 | 6
ASA Class [Number; unit: participants] — American Society of Anesthesiologists: ASA physical status classification system to assess fitness of patients before surgery.
  Classifications range from 1 (Healthy Person) to 6 (Declared brain-dead)
  Only participants in groups 1 and 2 (Healthy or mild systemic disease) are eligible to become living kidney donors.
  participants
    1 | 9 | 17 | 26
    2 | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Use (mg)
Description: Total Morphine Equivalents - mean in mg
Time Frame: Intra-Operative on day of surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
mg | 113.8 (19) | 99.6 (25)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Narcotic Use (mg)
Description: Total Morphine Equivalents - mean in mg
Time Frame: Post-operative (until time of discharge, typically 2-4 days)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
mg | 130.8 (125.6) | 134.5 (80.2)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.92, t-test, 2 sided

3. Primary Outcome: Narcotic Use (mg)
Description: Total Morphine Equivalent - mean in mg
Time Frame: Operative and Post-operative (until time of discharge, typically 2-4 days)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
mg | 244.6 (126.7) | 234.0 (88.0)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.78, t-test, 2 sided

4. Secondary Outcome: Subjective Pain Score
Description: Pain assessment via Visual Analogue Scale (VAS). Patients indicate pain on a continuous line which converts to a measured value in centimeters (cm). (Range: 0.0 and 10.0) - A score of 0 indicates no pain.
Time Frame: 1 hour post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
units on a scale | 4.6 (3.2) | 5.3 (3.2)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.52, t-test, 2 sided

5. Secondary Outcome: Subjective Pain Score
Description: Pain assessment via Visual Analogue Scale (VAS). Patients indicate pain on a continuous line which converts to a measured value in centimeters (cm). (Range: 0.0 and 10.0)- A score of 0 indicates no pain.
Time Frame: 6 hours post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
units on a scale | 3.5 (3.2) | 4.6 (2.6)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.25, t-test, 2 sided

6. Secondary Outcome: Subjective Pain Score
Description: as for outcome 4
Time Frame: 12 hours post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
units on a scale | 3.9 (3.0) | 3.7 (2.7)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.82, t-test, 2 sided

7. Secondary Outcome: Mean ETCO2
Description: mean End-tidal carbon dioxide concentration in the expired air
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Number analyzed (Participants) | 14 | 27
mmHg | 29.7 (4.4) | 30.8 (3.0)
Statistical Analysis 1: Comparison: Conventional Pressure vs Low Pressure (VTI); Test type: Superiority or Other; p = 0.45, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Description: Systematic chart reviews were conducted
Arm/Group | Conventional Pressure | Low Pressure (VTI)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/27
Other Adverse Events (participants affected / at risk) | 3/14 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Pressure (N=14) | Low Pressure (VTI) (N=27)
Post-operative hemorrhage (Surgical and medical procedures) | 1 (1) | 0 (0)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less